CLINICAL TRIAL: NCT06784544
Title: The Effects of Repeated Operational Stress and Limited Recovery on Resilience Capacity
Acronym: REP DEF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Collaborators: Pennington Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 24-33HC; MO240019 (Other Grant/Funding Number: Military Operational Medicine Research Program)
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Sleep, Inadequate; Energy Deficit; Iron Absorption; High Physical Activity
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: Randomized, parallel arm study. All volunteers will complete a 48h energy balance phase preceding two repeated rounds of 72h energy deficit (increased physical activity and reduced dietary intake) with sleep restriction (4h sleep opportunity / night) followed by a 48h recovery phase (energy balance, no physical activity, 7-9h sleep opportunity / night).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active adults representative of overweight phenotype (Experimental): Active adults representative of overweight phenotype will complete a 48h balance phase followed by two rounds of repeated 72h energy deficit exposure, each immediately followed by a 48h recovery phase.
  Interventions: Other: Operational Stressors
- Active adults representative of normal weight phenotype (Active Comparator): Active adults representative of normal weight phenotype will complete a 48h balance phase followed by two rounds of repeated 72h energy deficit exposure, each immediately followed by a 48h recovery phase.
  Interventions: Other: Operational Stressors

INTERVENTIONS:
Other: Operational Stressors — Intervention consists of a 48 hour energy balance phase preceding two rounds of repeated 72 hour energy deficit exposure each immediately followed by a 48h recovery phase. Balance and recovery phases will meet 100% of baseline energy requirements. Energy deficit phases will include an approximate 60% energy deficit of total daily energy requirements achieved through both a reduction in dietary intake and increased energy expenditure through physical activity.

SUMMARY:
This longitudinal study will examine the effects of repeated bouts of operational stress and limited recovery on integrated MPS, whole-body protein balance, iron absorption, and aerobic performance. Following baseline characterization measures, active adults (n=24) representative of normal weight phenotype (NW; n=12) and overweight phenotype (OW; n=12) will complete a 48h balance phase preceding two rounds of repeated 72h energy deficit exposure each immediately followed by a 48h recovery phase. NW cutoff will be defined ≤ 22% body fat for males and ≤ 32% body fat for females. OW cutoff will be defined as >22% body fat for males and >32% body fat for females. These body composition cutoffs are informed by the maximum allowable percent body fat standards outlined in current Army Regulation 600-9. Additional details for determining % body fat are outlined in the experimental procedures section of the protocol.

DETAILED DESCRIPTION:
Operational stress inherent of military training and operations is largely unavoidable and jeopardizes Warfighter readiness and performance. Operational stressors, including high physical activity, severe energy deficiency, and restricted sleep, challenge Warfighter resilience. The characterization of physiological factors contributing to maintained or declining resilience during repeated stress exposures with limited recovery is therefore required to enable development of new, targeted interventions that maintain or enhance resilience. Previous efforts have characterized the regulation of physiological status, including muscle recovery and endocrine function, during operational stress. However, no studies have directly assessed the effects of limited recovery (i.e., 48h) on physiological and performance decrements associated with repeated operational stress or resilience capacity. It is possible that repeated missions and limited recovery will drive progressive declines of physiological status and performance. The effects of operational stress on nutrition status also negatively impact readiness and performance. Absorption of key dietary nutrients, such as iron, is required to sustain nutritional status; and iron status, specifically, has been associated with performance declines. Laboratory and field-based studies from our group have shown declines in iron status and absorption following a single simulated sustained operation. However, no studies have directly assessed the effects of limited recovery (i.e., 48h) on physiological and performance decrements associated with repeated operational stress or resilience capacity. It is possible that repeated missions and limited recovery will drive progressive declines of physiological status and performance. Beyond characterizing the effects of repeated cycles of operational stress, there is potential value in determining whether body composition phenotypes (i.e., "energy deficiency-sensitive" and "energy deficiency-resistant") may modulate resilience during energy deficiency. Should phenotype-based differences be determined and suggest more beneficial/resilient vs. less beneficial/less resilient body composition phenotypes, guidance to maintain or interventions to achieve optimal body composition are potential individualized strategies to enhance resilience.

This longitudinal study will examine the effects of repeated operational stress and limited recovery on integrated muscle protein synthesis, whole-body protein balance, iron absorption, and aerobic performance. Adults (n=24) representative of normal weight and overweight phenotype (n=12/phenotype) will complete a 48h balance phase preceding two repeated rounds of 72h energy deficit (increased physical activity and reduced dietary intake) with sleep restriction followed by a 48h recovery phase.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 - 39 years (17 - 39 years if military personnel)
* Weight stable in the past 2 months (± approximately 5 kg)
* Healthy without evidence of chronic illness or musculoskeletal injury as determined by the USARIEM Office of Medical Support and Oversight (OMSO) or home duty station medical support (HMS)
* Functional exercise (i.e., step ups, box jumps, body mass movements) and/or aerobic exercise trained defined by self-report as performing ≥ 2 sessions/wk for previous 6 months
* Willing to refrain from alcohol, smoking any nicotine product (includes e-cigarettes); vaping, chewing tobacco, caffeine not provided in the study, and dietary supplement use throughout the dietary interventions
* Biological females must be on sustained (i.e., approximately >3 months) oral/hormonal contraceptive use which acts to maintain continuous hormonal levels (i.e., contains low-dose estrogen/progesterone with no oral placebos, hormonal IUD)
* Supervisor approval for federal civilian employees and non-HRV active duty military personnel)

Exclusion Criteria:

* Musculoskeletal injuries that compromise exercise capability as determined by OMSO or HMS
* Metabolic or cardiovascular abnormalities, sleep disorders (i.e., sleep apnea) gastrointestinal disorders (e.g., kidney disease, diabetes, cardiovascular disease, etc.) as determined by OMSO or HMS
* Abnormal or problems with blood clotting as determined by OMSO or HMS
* History of complications with lidocaine or similar local anesthetic analogue
* Present condition of alcoholism, anabolic steroids, or other substance abuse issues
* Blood donation within 8-wk of beginning or completing study blood draws
* Current diagnosis of Anemia (hemoglobin < 13 g/dL for males, hemoglobin < 12 g/dL for females) and Sickle Cell Anemia/Trait as determined by OMSO or HMS
* Pregnant, trying to become pregnant, and/or breastfeeding (results of urine pregnancy test or self-report for breastfeeding will be obtained before body composition testing)
* Claustrophobia or discomfort related to having enclosed equipment around the head
* Unwillingness or inability to consume study diets or foods provided due to personal preference or food allergies/sensitivities
* Unwillingness or inability to adhere to study exercise restrictions and prescriptions

Ages: 17 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Integrated muscle protein synthesis | Days 1-13
  deuterium oxide stable isotope
Whole-body protein balance | 24 hours
  15N alanine stable isotope
Iron Absorption | 24 hours
  57-Fe dissolved in water

CONTACTS AND LOCATIONS:
Overall Officials: Jess A Gwin Principal Investigator, PhD, Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- US Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.